CLINICAL TRIAL: NCT00697411
Title: Pathogenesis of Selected X-Linked Dominant Disorders and New Strategies to Identify the Gene Mutated in Aicardi Syndrome
Brief Title: Study of Selected X-Linked Disorders: Aicardi Syndrome
Status: Recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: Aicardi Syndrome Foundation (Other)
Responsible Party: Principal Investigator, Ignatia Van den Veyver, Professor, Baylor College of Medicine
Other Study IDs: BCM Aicardi H12791
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Aicardi Syndrome; Brain Disorders
Keywords: Aicardi syndrome; Neurodevelopmental disorders; X-linked disorders
MeSH Terms: conditions — Aicardi Syndrome; Brain Diseases; Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — lymphoblast DNA; tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Individuals with Aicardi syndrome and their first-degree relatives
  Interventions: Other: Syndrome cause identification

INTERVENTIONS:
Other: Syndrome cause identification

SUMMARY:
Based on our current understanding of Aicardi syndrome, the condition is hypothesized to occur due to a genetic change on the X-chromosome. The research team is investigating Aicardi syndrome to identify the specific gene location associated with the disorder. The investigators are collecting blood and skin biopsy samples from patients and their parents. A permanent cell line is prepared and DNA from the blood and skin samples and cell lines is isolated and then used for genetic testing. The current research includes microarray analysis which which is used to look for duplications or deletions of genetic material, mutation analysis of candidate genes by sequencing, genome-wide sequencing, review of medical records to identify trends suggesting possible candidate genes of interest, and X chromosome inactivation studies.

DETAILED DESCRIPTION:
Aicardi syndrome is a sporadic X-linked dominant, presumably male-lethal, neurodevelopmental disorder. It was initially characterized by agenesis of the corpus callosum, neuronal migration defects, eye abnormalities (chorioretinal lacunae, colobomas of the optic nerve and microphthalmia) and severe early-onset seizures and neurodevelopmental delay. It is now well recognized that other brain abnormalities, such as polymicrogyria, agyria, cysts and heterotopias are common features of Aicardi syndrome. The investigators previously hypothesized that the gene causing Aicardi syndrome and possibly additional phenotypically similar disorders with X-linked inheritance, such as Goltz syndrome or Focal Dermal Hypoplasia, are in or near the region on chromosome Xp22 that is deleted in another condition named microphthalmia with linear skin defects syndrome (MLS), because all three have some clinical similarities. However, interim studies have shown that this is likely not the case because no mutations were found in Aicardi syndrome in human holocytochrome c-type synthetase (HCCS) , the gene that is deleted or mutated in MLS. In addition, a mouse model for MLS has no features of Aicardi syndrome. Furthermore, the ivnestigators identified mutations in PORCN (Xp11.3) in Goltz syndrome patients, but not in Aicardi syndrome patients. Therefore, it is likely that the mutated gene is elsewhere on the X-chromosome.

For this study the investigators are collecting information on patients with clinical findings suggesting a diagnosis of Aicardi syndrome, MLS syndrome or a condition that phenotypically overlaps with these disorders. A detailed family history will be obtained, when indicated, and additional family members will be evaluated after appropriately obtained written voluntary consent. A detailed report of the history or physical findings will be obtained from referring physicians for patients identified at outside facilities, or the participants may be evaluated by the study collaborators. Blood and skin biopsy will be obtained from affected individuals, unaffected parents and from other affected or unaffected family members where indicated. It is anticipated that some severely affected patients will expire; in that case, (post mortem) pathological specimens may be obtained. Occasionally, affected individuals may undergo surgical procedures with removal of tissues; in this case we may obtain tissues that would be otherwise discarded or that are not essential for further diagnostic studies or clinical care of the patient. It is anticipated that these specimens will be extremely valuable for understanding the pathogenesis of the investigated conditions. DNA, RNA or protein will be prepared from leukocytes and from tissues and used for sequencing and mutation analysis and other molecular studies of the identified genes. Permanent lymphoblastoid cell lines will be prepared and stored in the laboratory as a permanent source of DNA for the molecular studies. Cell lines may be made from skin biopsies

ELIGIBILITY:
Inclusion Criteria:

* Features suggestive of Aicardi syndrome (not all features must be present)

  * Agenesis of the corpus callosum
  * Chorioretinal lacunae
  * Seizures (infantile spasms)

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Girls with Aicardi syndrome and their unaffected parents. Sometimes additional family members are also enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2002-10 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Identifying the change in the genetic information that causes Aicardi syndrome | Through study completion, an average of 20 years
  The investigators will isolate genetic material from samples of individuals with Aicardi syndrome and their parents (if available). DNA sequencing and other molecular methods along with bioinformatic analysis will be used to find genetic variants (changes) in the genetic code unique to individuals with Aicardi syndrome, not seen in healthy population. When a gene that shows variants that are deleterious to its function is identified in at least 3 unrelated Aicardi syndrome individuals but not in healthy people (whose DNA sequence is in public databases), the outcome (finding the genetic cause of Aicardi syndrome) will be achieved. Aicardi syndrome is very rare, thus recruitment and enrollment of new individuals will continue when they are referred to the study. In this research a key finding in one individual can provide the clue for the entire cohort. It cannot be predicted when this will happen, thus enrollment and data collection will continue as long as the study is ongoing.

CONTACTS AND LOCATIONS:
Overall Officials: Ignatia B Van den Veyver, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient data with all identification removed will be published following peer review in journals and/or presented at scientific meetings.
Time Frame: At the end of the study.
Access Criteria: Patient data with all identification removed will be published following peer review in journals and/or presented at scientific meetings.
  Reasonable requests from other researchers working on the same disease will be reviewed by the PI and sharing will be done after full deidentification and with institutionally approved of data and material transfer agreements.

REFERENCES:
- [Background] Aicardi, J, Levebre, J, and Lerique-Koechlin, A (1965) A new syndrome: Spasms in flexion, callosal agenesis, ocular abnormalities. Electroencephalogr Clin Neurophysiol 19, 609-610.
- [Background] Donnenfeld AE, Packer RJ, Zackai EH, Chee CM, Sellinger B, Emanuel BS. Clinical, cytogenetic, and pedigree findings in 18 cases of Aicardi syndrome. Am J Med Genet. 1989 Apr;32(4):461-7. doi: 10.1002/ajmg.1320320405. PMID 2773986
- [Background] Kitamura K, Yanazawa M, Sugiyama N, Miura H, Iizuka-Kogo A, Kusaka M, Omichi K, Suzuki R, Kato-Fukui Y, Kamiirisa K, Matsuo M, Kamijo S, Kasahara M, Yoshioka H, Ogata T, Fukuda T, Kondo I, Kato M, Dobyns WB, Yokoyama M, Morohashi K. Mutation of ARX causes abnormal development of forebrain and testes in mice and X-linked lissencephaly with abnormal genitalia in humans. Nat Genet. 2002 Nov;32(3):359-69. doi: 10.1038/ng1009. Epub 2002 Oct 15. PMID 12379852
- [Background] Prakash SK, Cormier TA, McCall AE, Garcia JJ, Sierra R, Haupt B, Zoghbi HY, Van Den Veyver IB. Loss of holocytochrome c-type synthetase causes the male lethality of X-linked dominant microphthalmia with linear skin defects (MLS) syndrome. Hum Mol Genet. 2002 Dec 1;11(25):3237-48. doi: 10.1093/hmg/11.25.3237. PMID 12444108
- [Background] Schaefer L, Ballabio A, Zoghbi HY. Cloning and characterization of a putative human holocytochrome c-type synthetase gene (HCCS) isolated from the critical region for microphthalmia with linear skin defects (MLS). Genomics. 1996 Jun 1;34(2):166-72. doi: 10.1006/geno.1996.0261. PMID 8661044
- [Background] Schaefer L, Prakash S, Zoghbi HY. Cloning and characterization of a novel rho-type GTPase-activating protein gene (ARHGAP6) from the critical region for microphthalmia with linear skin defects. Genomics. 1997 Dec 1;46(2):268-77. doi: 10.1006/geno.1997.5040. PMID 9417914
- [Background] Stromme P, Mangelsdorf ME, Scheffer IE, Gecz J. Infantile spasms, dystonia, and other X-linked phenotypes caused by mutations in Aristaless related homeobox gene, ARX. Brain Dev. 2002 Aug;24(5):266-8. doi: 10.1016/s0387-7604(02)00079-7. PMID 12142061
- [Background] Van den Veyver IB. Microphthalmia with linear skin defects (MLS), Aicardi, and Goltz syndromes: are they related X-linked dominant male-lethal disorders? Cytogenet Genome Res. 2002;99(1-4):289-96. doi: 10.1159/000071606. PMID 12900577
- [Background] Van den Veyver IB, Cormier TA, Jurecic V, Baldini A, Zoghbi HY. Characterization and physical mapping in human and mouse of a novel RING finger gene in Xp22. Genomics. 1998 Jul 15;51(2):251-61. doi: 10.1006/geno.1998.5350. PMID 9722948
- [Result] Zhang W, Amir R, Stockton DW, Van Den Veyver IB, Bacino CA, Zoghbi HY. Terminal osseous dysplasia with pigmentary defects maps to human chromosome Xq27.3-xqter. Am J Hum Genet. 2000 Apr;66(4):1461-4. doi: 10.1086/302868. Epub 2000 Mar 17. PMID 10739772
- [Result] Sutton VR, Hopkins BJ, Eble TN, Gambhir N, Lewis RA, Van den Veyver IB. Facial and physical features of Aicardi syndrome: infants to teenagers. Am J Med Genet A. 2005 Oct 15;138A(3):254-8. doi: 10.1002/ajmg.a.30963. PMID 16158440
- [Result] Glasmacher MA, Sutton VR, Hopkins B, Eble T, Lewis RA, Park Parsons D, Van den Veyver IB. Phenotype and management of Aicardi syndrome: new findings from a survey of 69 children. J Child Neurol. 2007 Feb;22(2):176-84. doi: 10.1177/0883073807300298. PMID 17621479
- [Result] Wang X, Reid Sutton V, Omar Peraza-Llanes J, Yu Z, Rosetta R, Kou YC, Eble TN, Patel A, Thaller C, Fang P, Van den Veyver IB. Mutations in X-linked PORCN, a putative regulator of Wnt signaling, cause focal dermal hypoplasia. Nat Genet. 2007 Jul;39(7):836-8. doi: 10.1038/ng2057. Epub 2007 Jun 3. PMID 17546030
- [Result] Fruhman G, Eble TN, Gambhir N, Sutton VR, Van den Veyver IB, Lewis RA. Ophthalmologic findings in Aicardi syndrome. J AAPOS. 2012 Jun;16(3):238-41. doi: 10.1016/j.jaapos.2012.01.008. PMID 22681940
- [Result] Wang X, Sutton VR, Eble TN, Lewis RA, Gunaratne P, Patel A, Van den Veyver IB. A genome-wide screen for copy number alterations in Aicardi syndrome. Am J Med Genet A. 2009 Oct;149A(10):2113-21. doi: 10.1002/ajmg.a.32976. PMID 19760649
- [Result] Eble TN, Sutton VR, Sangi-Haghpeykar H, Wang X, Jin W, Lewis RA, Fang P, Van den Veyver IB. Non-random X chromosome inactivation in Aicardi syndrome. Hum Genet. 2009 Mar;125(2):211-6. doi: 10.1007/s00439-008-0615-4. Epub 2009 Jan 1. PMID 19116729
- [Result] Hopkins B, Sutton VR, Lewis RA, Van den Veyver I, Clark G. Neuroimaging aspects of Aicardi syndrome. Am J Med Genet A. 2008 Nov 15;146A(22):2871-8. doi: 10.1002/ajmg.a.32537. PMID 18925666
- [Result] Van den Veyver IB, Panichkul PP, Antalffy BA, Sun Y, Hunter JV, Armstrong DD. Presence of filamin in the astrocytic inclusions of Aicardi syndrome. Pediatr Neurol. 2004 Jan;30(1):7-15. doi: 10.1016/s0887-8994(03)00311-4. PMID 14738943
- [Result] Wong BK, Sutton VR, Lewis RA, Van den Veyver IB. Independent variant analysis of TEAD1 and OCEL1 in 38 Aicardi syndrome patients. Mol Genet Genomic Med. 2017 Jan 25;5(2):117-121. doi: 10.1002/mgg3.250. eCollection 2017 Mar. PMID 28361097